CLINICAL TRIAL: NCT05438420
Title: A Phase 1B/2, Open-label Study of Q702 in Combination With Intravenous Pembrolizumab in Patients With Selected Advanced Solid Tumors
Brief Title: Oral Axl/Mer/CSF1R Selective Tyrosine Kinase Inhibitor Q702 in Combination With Pembrolizumab in Patients With Selected Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qurient Co., Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QRNT-008; MK-3475-D35 (KEYNOTE-D35) (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2022-05-20; First posted 2022-06-30 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Cancer; Gastric Cancer; Hepatocellular Cancer; Cervical Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Liver Neoplasms; Uterine Cervical Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation of Q702 in combination with fixed dose of pembrolizumab (Experimental): Give one week on/one week off at selected dose level
  Interventions: Drug: Q702; Biological: Pembrolizumab
- Dose expansion of Q702 in combination with fixed dose of pembrolizumab (Experimental): Give intravenously once every three week at 200 mg
  Interventions: Drug: Q702; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Q702 — The study drug Q702 will be administered once daily by mouth on Days 1 through 7, Days 15 through 21 and Days 29 through 35 of every treatment cycle.
Biological: Pembrolizumab — Pembrolizumab will be administered using IV infusion on Day 1 of each 3-week treatment cycle
  Other Names: KEYTRUDA®

SUMMARY:
This study is a phase 1B/2 open-label, study to determine safety and preliminary efficacy of Q702 in combination with pembrolizumab in study subjects with advanced esophageal, gastric/GEJ, hepatocellular, and cervical cancers.

ELIGIBILITY:
Inclusion Criteria:

* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Subjects with histologically or cytologically confirmed advanced or metastatic esophageal, gastric/GEJ, hepatocellular and cervical cancers who have progressed on treatment with an anti-PD1 or anti PD-L1 monoclonal antibody (mAb) administered either as monotherapy, or in combination with other therapies
* Have measurable disease per RECIST v 1.1. as assessed by local site investigator/radiology
* Have an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy of at least 3 months

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test (within 72 hours) prior to treatment or breast-feeding women
* Concomitant use of strong inhibitors and inducers of CYP1A2, 2J2, 2C19, 2D6, and 3A4/5 within the timeline duration of five half-lives prior to starting study drug and throughout the trial
* Concomitant use of sensitive substrates of CYP2C9, 2C19, and 3A4 within the timeline duration of five half-lives prior to starting study drug and throughout the trial
* Has received prior radiotherapy within 2 weeks of start of study treatment or have had a history of radiation pneumonitis
* Has had an allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE | Up to approximately 2 years (Each Cycle is 42 Days)
Tumor response using RECIST version 1.1 throughout study | Up to approximately 2 years (Each Cycle is 42 Days)

SECONDARY OUTCOMES:
Change in the area under curve (AUC) of Q702 and its primary metabolites | Cycle 1 Day 1 and Day 22 (Each Cycle is 42 Days)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Norton Cancer Institute, Louisville, Kentucky
- South Korea (5):
  - CHA Bundang Medical Center, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided